CLINICAL TRIAL: NCT06810440
Title: Reducing Anemia Among Young Preconception Women in Nepal Through a Group Household Norm and Micronutrient Supplementation Intervention
Brief Title: Reducing Anemia Among Preconception Women in Nepal Through a Group Norm and Micronutrient Supplementation Intervention
Acronym: Sumadhur
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Center for Research on Environment, Health and Population Activities (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD114798 (NIH); R01HD114798 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Anemia, Iron-Deficiency; Nutritional Deficiencies; Adherence; Norms, Social; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Anemia, Iron-Deficiency; Malnutrition; Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm will receive the standard of care and the intervention at the end of the study period
- Intervention (Experimental): Sumadhur is a 4-month intervention with weekly sessions that last about 1.5 hours. Newly married women, their husbands and mothers-in-law gather with other household triads (5 households per group for a total of 15 people per group). Intervention participants will also receive multiple micronutritent supplements (MMS)
  Interventions: Behavioral: Sumadhur; Dietary Supplement: Multiple micronutrient supplement MMS

INTERVENTIONS:
Behavioral: Sumadhur — Sumadhur is a 4-month intervention with weekly sessions that last about 1.5 hours. Newly married women, their husbands and mothers-in-law gather with other household triads (5 households per group for a total of 15 people per group).
  Arms: Intervention
Dietary Supplement: Multiple micronutrient supplement MMS — Multiple micronutrient supplement MMS provided in 180 pill bottles
  Arms: Intervention

SUMMARY:
Preconception micronutrient status (including anemia) is a critical determinant of maternal, newborn, and child health that remains undervalued in Nepal. However, providing micronutrient supplements (MMS) alone is not enough. In the Nepali context, the gap between marriage and the first birth is short and newly married women have the lowest household status. Addressing the intersectional barriers to health for newly married women, including inequitable gender norms and women's empowerment, household relationships, nutrition knowledge and practices-is essential for improving maternal and infant outcomes in Nepal. To mitigate the community, household, and individual factors resulting in poor nutrition, the team developed and pilot-tested an educational group intervention (Sumadhur, meaning "Best Relationship") for newly married women, husbands, and mothers-in-law triads. Sumadhur aims to provide information on nutrition and women's health, address inequitable gender norms and practices, strengthen household relationships and communication, and improve the household status of newly married women. The pilot study of Sumadhur brought triads of several households together for 16 interrelated sessions over four-months. Findings suggest that participants (N=90) found the intervention to be highly feasible and acceptable and nutritional norms and practices improved.

We propose to test the effectiveness of Sumadhur on maternal health and nutrition outcomes using a 2-arm cluster RCT (cRCT). The intervention participants will receive the Sumadhur group intervention and will be provided MMS directly at group sessions. In control villages who do not receive the Sumadhur group intervention, we will facilitate access to MMS at primary health centers. We will randomize 70 villages to each arm (with one group per village). Each village has one group of five women (total of 700 women). Newly married women, their husbands and mothers-in-laws (total=2,100), will be followed four times for 18 months post-intervention through surveys, hemoglobin tests and blood draws (women only). The specific aims are to estimate the effectiveness of Sumadhur on women's anemia and micronutrient status, including the cost-benefit of the intervention (Aim 1); explore the impact on intermediate outcomes such as gender norms, household relationships and eating practices and characterize the individual and household-level mechanisms of impact (Aim 2); understand triadic experiences and impact over time of Sumadhur (Aim 3).

Accomplishing these aims will provide evidence for how to improve micronutrient and anemia status among women before they become pregnant-thereby ensuring that women are not deficient in the critical early phases of pregnancy. These findings will also advance the field by testing novel approaches (household and community level behavior and norm change intervention) that, when combined with supplements, may lead to better adherence, uptake, and, ultimately, health outcomes, and have additional longer-term benefits.

DETAILED DESCRIPTION:
Anemia and micronutrient (iron, folate, B12, zinc) deficiencies during pregnancy are a leading cause of maternal mortality and morbidity in South Asia and have intergenerational effects, contributing to low birth weight, preterm birth and perinatal mortality. Despite national efforts to provide iron-folic acid (IFA) supplements to pregnant women in Nepal for free, only 41% consume the recommended amount, and high levels of maternal anemia (52%) and micronutrient deficiencies persist. Provision of micronutrient supplements is necessary but not sufficient-intersectional social and behavioral factors also must be addressed. Furthermore, micronutrient status needs to be improved during the preconception period to impact the important first trimester (before most women in Nepal typically seek care) to improve maternal and infant outcomes to the greatest extent possible. With short gaps between marriage and first pregnancy, newly married women should be a focal population. National health and nutrition programs do not currently provide micronutrient supplementation (MMS) to preconception women nor do they mitigate the structural, social, and behavioral (ecological) factors.

Several barriers to adequate nutrition and potential uptake of MMS have been identified. Inequitable gender norms limit women's access to nutrition and health care in South Asia, where women, especially young and newly married, have low levels of empowerment. Women's limited agency in the household and community lead women to have poor dietary diversity, low consumption of micronutrient-rich foods and seek antenatal care late. Household food insecurity and incomplete nutrition knowledge also contribute to women's poor nutritional status preconception and in pregnancy. Hence, engaging other household members (husbands and in-laws) and addressing broader issues around women's status are key to reducing anemia and improving micronutrient status. To address these barriers, interventions engaging multiple household members are necessary to shift norms and promote healthy behavior change, in addition to providing information and access to MMS. Formative research in rural Nepal (K01HD086281) found that newly married women, their husbands, and mothers-in-law ("triads") desired information about nutrition and maternal health. Investigators found that young (<25 years) newly married women often ate last and had low dietary diversity, and positive household relationships were associated with enhanced access to nutritious foods. Thus, in collaboration with local community partners, the investigators developed Sumadhur, a 4-month group intervention that covers preconception and pregnancy nutrition, household eating patterns, anemia, maternal healthcare seeking, gender norms and inequality, and couples/household relationship dynamics. Triads met weekly with other triads (5 households per group=15 people per group). Pilot data from six groups (N=90 participants) found Sumadhur to be acceptable and feasible (83% attended >80% of sessions) and showed preliminary evidence of changes in nutrition norms and practices.8 Based on these promising preliminary findings, the investigators propose to test the effectiveness of Sumadhur on maternal health and nutrition outcomes using a 2-arm cluster randomized controlled trial. Intervention participants will receive the Sumadhur group intervention and be provided MMS directly at group sessions whereas MMS will be freely available at primary health centers in control villages. The investigators will randomize 70 villages to each arm (140 villages total). Each village will have one group of ~5 newly married women, their husbands and mothers-in-laws (N=2,100), who will be followed every 4-6 months for 18-months post-intervention through surveys, hemoglobin assessments and blood draws (women only). The investigators will conduct concurrent in-depth longitudinal qualitative interviews (LQIs) with a sub-set of triads at each data collection time points.

Aim 1: To estimate the effectiveness of Sumadhur on newly married women's anemia and micronutrient deficiency. The primary effectiveness outcomes are the prevalence of anemia (hemoglobin <12g/dL or <11g/dL if pregnant) and deficiencies/insufficiencies in selected micronutrients: iron, zinc, vitamin B12, and folate (1a).

Secondary outcomes include reproductive, pregnancy/maternal and infant health behaviors and outcomes. The investigators will also determine the cost per disability-adjusted life year averted of the intervention to inform scale-up (1b).

Aim 2: To estimate the (a) effectiveness and (b) mechanism of impact of Sumadhur on intermediary outcomes that may be on the causal path to improved anemia and micronutrient status. The primary outcomes for aim 2a are: (1) social and gender norms, (2) women's empowerment, (3) nutrition and maternal health knowledge, and (4) household relationships and eating patterns, using data collected from all members of triads. In 2b, the investigators will delineate the pathways through which Sumadhur operates, including changing intermediary outcomes and MMS adherence using mediation analyses to identify drivers of intervention impact.

Aim 3: Understand triadic experiences and impact over time of Sumadhur. Using a convergent parallel analysis design, the investigators will uncover explanations for these quantitative findings from multiple perspectives using triadic longitudinal IDI data from newly married women, their husbands, and mothers-in-law.

The investigators' findings will inform programs and policies aiming to reduce anemia and micronutrient deficiencies, which are key contributors to excess maternal, newborn, and child morbidity and mortality globally. This work will lay the groundwork for potential implementation studies of the scale-up and integration into Nepal's National Policy.

ELIGIBILITY:
Inclusion Criteria:

* the newly married couple having been married in the last four months
* women being under 25 years old
* never pregnant and not currently pregnant
* co-residing with the mother-in-law in a household as defined by sharing meals together.
* all triad-household members must also be willing to participate
* husbands must not be planning to migrate in the next 6 months.

Exclusion Criteria:

* Over 25, under 18 years old
* Currently or ever pregnant
* married more than 4 months before
* not co-residing
* not being willing to participate.
* do not consent to blood-draws
* women who are severely anemic (hemoglobin < 8.0 g/dL) at baseline based on hemoglobin via Hemocue assessment of a fingerprick blood sample at the time of enrollment

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Participants with Anemia | 6 months
  Participants with hemoglobin <12g/dL or <11g/dL if pregnant will be considered anemic
Participants with deficiencies/insufficiencies in selected micronutrients | 6 months
  Participants with deficiencies in the following micronutrients: iron, vitamin B12, and folate

SECONDARY OUTCOMES:
Body max index | 18 months
  Body Mass Index measured with weight in kilograms over height in cm
Pregnancy status | 18 months
  Self reported pregnancy, measured using date of last menstrual period

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for Research on Environment, Health and Population Activities (CREHPA), Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keats EC, Haider BA, Tam E, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2019 Mar 14;3(3):CD004905. doi: 10.1002/14651858.CD004905.pub6. PMID 30873598
- [Background] Bourassa MW, Osendarp SJM, Adu-Afarwuah S, Ahmed S, Ajello C, Bergeron G, Black R, Christian P, Cousens S, de Pee S, Dewey KG, Arifeen SE, Engle-Stone R, Fleet A, Gernand AD, Hoddinott J, Klemm R, Kraemer K, Kupka R, McLean E, Moore SE, Neufeld LM, Persson LA, Rasmussen KM, Shankar AH, Smith E, Sudfeld CR, Udomkesmalee E, Vosti SA. Review of the evidence regarding the use of antenatal multiple micronutrient supplementation in low- and middle-income countries. Ann N Y Acad Sci. 2019 May;1444(1):6-21. doi: 10.1111/nyas.14121. Epub 2019 May 27. PMID 31134643
- [Background] Morrison J, Giri R, Arjyal A, Kharel C, Harris-Fry H, James P, Baral S, Saville N, Hillman S. Addressing anaemia in pregnancy in rural plains Nepal: A qualitative, formative study. Matern Child Nutr. 2021 Jul;17 Suppl 1(Suppl 1):e13170. doi: 10.1111/mcn.13170. PMID 34241951
- [Background] Daru J, Zamora J, Fernandez-Felix BM, Vogel J, Oladapo OT, Morisaki N, Tuncalp O, Torloni MR, Mittal S, Jayaratne K, Lumbiganon P, Togoobaatar G, Thangaratinam S, Khan KS. Risk of maternal mortality in women with severe anaemia during pregnancy and post partum: a multilevel analysis. Lancet Glob Health. 2018 May;6(5):e548-e554. doi: 10.1016/S2214-109X(18)30078-0. Epub 2018 Mar 20. PMID 29571592
- [Background] Rahman MM, Abe SK, Rahman MS, Kanda M, Narita S, Bilano V, Ota E, Gilmour S, Shibuya K. Maternal anemia and risk of adverse birth and health outcomes in low- and middle-income countries: systematic review and meta-analysis. Am J Clin Nutr. 2016 Feb;103(2):495-504. doi: 10.3945/ajcn.115.107896. Epub 2016 Jan 6. PMID 26739036
- [Derived] Diamond-Smith N, Puri MC, Borak L, Walker D, Charlebois E, Weiser SD, McDonald CM. Cluster randomised controlled trial of a household-level, group preconception nutrition awareness and norm intervention (SUMADHUR) combined with multiple micronutrient supplements (MMS) for newly married households: a protocol. BMJ Open. 2025 Jul 25;15(7):e103488. doi: 10.1136/bmjopen-2025-103488. PMID 40713050